CLINICAL TRIAL: NCT00248521
Title: A Cancer Research UK Phase I Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of 17-Dimethylaminoethyl-amino-17-Demethoxygeldanamycin (17-DMAG) Given as a Once Weekly Infusion in Patients With Advanced Solid Tumors
Brief Title: 17-Dimethylaminoethylamino-17-Demethoxygeldanamycin (17-DMAG) in Treating Patients With Metastatic Solid Tumors or Tumors That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ICR-PH1/102; CDR0000442402 (Registry Identifier: PDQ (Physician Data Query)); NCI-6547
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: alvespimycin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG), work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-DMAG in treating patients with metastatic solid tumors or tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose, dose-limiting toxicity, and recommended phase II dose of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) in patients with unresectable or metastatic solid tumors.
* Determine the feasibility, safety, and toxicity profile of this drug in these patients.

Secondary

* Determine the clinical pharmacokinetic profile of this drug in these patients.
* Determine tumor response in patients treated with this drug.
* Determine the biologically effective dose.

OUTLINE: This is an open-label, non-randomized, dose-escalation, multicenter study.

Patients receive 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) IV over 1 hour on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 17-DMAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD.

After completion of study treatment, patients are followed for 28 days.

PROJECTED ACCRUAL: Approximately 25-35 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor

  * Unresectable or metastatic disease
* Standard curative or palliative measures do not exist OR are no longer effective OR patient refused such measures
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin normal
* ALT and AST ≤ 1.5 times upper limit of normal
* No chronic liver disease
* Hepatitis B or C negative

Renal

* Creatinine normal OR
* Creatinine clearance normal

Cardiovascular

* No symptomatic New York Heart Association class III-IV cardiac disease
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No poorly controlled angina
* No uncontrolled dysrhythmia or dysrhythmias requiring antiarrhythmic drugs
* No transient ischemic attack
* No stroke
* No peripheral vascular disease
* No congenital long QT syndrome
* No history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* QTc < 450 msec (for men) and 470 msec (for woman)
* LVEF > 40% by MUGA
* No left bundle branch block

Pulmonary

* No symptomatic pulmonary disease requiring medication, including any of the following:

  * Dyspnea with or without exertion
  * Paroxysmal nocturnal dyspnea
  * Oxygen requirement
  * Significant pulmonary disease (e.g., chronic obstructive/restrictive pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks before, during, and for 6 months after completion of study treatment
* No known HIV positivity
* No other malignancy within the past 5 years except adequately treated cone biopsied carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No ongoing or active infection
* No diabetes mellitus (with evidence of severe peripheral vascular disease or ulcers)
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* Concurrent epoetin alfa allowed

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)

Endocrine therapy

* More than 4 weeks since prior endocrine therapy
* Concurrent luteinizing hormone-releasing hormone analogues for androgen-insensitive prostate cancer and rising prostate-specific antigen allowed

Radiotherapy

* More than 4 weeks since prior radiotherapy (except for palliative treatment)
* No prior irradiation field that potentially included the heart (e.g., mantle)

Surgery

* Not specified

Other

* Recovered from all prior therapy
* Concurrent bisphosphonates allowed
* At least 5 half-lives since prior and no concurrent medication that prolong QTc
* No other concurrent anticancer or investigational agents
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) at 28 days after treatment

SECONDARY OUTCOMES:
Heat shock protein 90 (HSP90) client protein and co-chaperone changes up to 29 days after treatment
Tumor response by RECIST criteria every 6 weeks while on study
Clinical pharmacokinetic profile established during the first course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ian R. Judson, MA, MD, FRCP, Study Chair — Institute of Cancer Research, United Kingdom
Locations (3):
- United Kingdom (3):
  - Institute of Cancer Research - Sutton, Sutton, England
  - Royal Marsden - Surrey, Sutton, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland

REFERENCES:
- [Result] Pacey SC, Wilson RH, Walton M, et al.: A phase I trial of the heat shock protein 90 (HSP90) inhibitor alvespimycin (17-dimethylaminoethylamino-17-demethoxygeldanamycin 17-DMAG) administered weekly, intravenously, to patients with advanced solid tumors. [Abstract] American Association for Cancer Research: Molecular Targets and Cancer Therapeutics, October 22-26, 2007, San Francisco, CA A-PR-6, 2007.